CLINICAL TRIAL: NCT02997254
Title: COMparison of Physiological Algorithms for Real-time Evaluation of Atrial Fibrillation
Acronym: COMPARE_AF
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sanjiv Narayan, MD, PhD, Professor of Medicine, Principal Investigator, Stanford University
Other Study IDs: COMPARE_AF
Record Dates: First submitted 2016-12-12; First posted 2016-12-20 (Estimated); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation; Abnormal Heart Rhythms
Keywords: atrial fibrillation; ablation; abnormal heart rhythm
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cohort study to evaluate algorithms for mapping atrial fibrillation by mapping atrial structure and mapping electrical activity to detect physiologically important areas.

A key innovation of the observation study is to assess tracking of physiological activity in AF, in relation to tissue activity (MAP recordings), and in relation to AF waves of activity.

This observational work extends prior studies that focused on focal and rotational activity, dispersion of electrical activity, low voltage activity and others.

DETAILED DESCRIPTION:
In this study, the investigators will compare mapping approaches for atrial fibrillation ablation.

First, investigators will compare approaches to map atrial structure from collected computed tomography (CT) scans or magnetic resonance imaging (MRI) scans acquired routinely in patients undergoing ablation for atrial fibrillation. Imaging will be acquired from a variety of clinically approved

Second, investigators will compare approaches to analyze electrograms collected routinely at clinical electrophysiology study (EPS) in patients undergoing ablation for atrial fibrillation. Electrograms will be recorded from a variety of clinically approved catheters under standard of care conditions, and will be analyzed to better understand the mechanisms for atrial fibrillation and its relationship to outcomes. Electrograms include unipolar recordings, bipolar recordings and, monophasic action potential recordings using FDA-cleared catheters.

The investigators anticipate analyzing data from 1000 patients from inception of the study.

ELIGIBILITY:
Inclusion Criteria:

* aged 21-80 yrs who underwent electrophysiology study for ablation of Atrial Fibrillation

Exclusion Criteria:

* Poor data quality of recordings of AF

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will study adults aged 21-90 years who have undergone electrophysiology study for ablation of Atrial Fibrillation. De-identified datasets will be made available for comparisons of mapping approaches.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy | At the time of procedure
  Comparing electrogram analysis systems to diagnose sites of importance in Atrial Fibrillation
Diagnostic Accuracy | At time of procedure.
  Comparing algorithms to segment atrial structures from computed tomography or Magnetic resonance images.

SECONDARY OUTCOMES:
Analysis Time | At time of procedure.
  Comparing time required to segment atrial structures from computed tomography or magnetic resonance images.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv M Narayan, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhusseini M, Vidmar D, Meckler GL, Kowalewski CA, Shenasa F, Wang PJ, Narayan SM, Rappel WJ. Two Independent Mapping Techniques Identify Rotational Activity Patterns at Sites of Local Termination During Persistent Atrial Fibrillation. J Cardiovasc Electrophysiol. 2017 Jun;28(6):615-622. doi: 10.1111/jce.13177. Epub 2017 Mar 20. PMID 28185348
- [Background] Alhusseini MI, Abuzaid F, Rogers AJ, Zaman JAB, Baykaner T, Clopton P, Bailis P, Zaharia M, Wang PJ, Rappel WJ, Narayan SM. Machine Learning to Classify Intracardiac Electrical Patterns During Atrial Fibrillation: Machine Learning of Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2020 Aug;13(8):e008160. doi: 10.1161/CIRCEP.119.008160. Epub 2020 Jul 6. PMID 32631100
- [Background] Tang S, Razeghi O, Kapoor R, Alhusseini MI, Fazal M, Rogers AJ, Rodrigo Bort M, Clopton P, Wang PJ, Rubin DL, Narayan SM, Baykaner T. Machine Learning-Enabled Multimodal Fusion of Intra-Atrial and Body Surface Signals in Prediction of Atrial Fibrillation Ablation Outcomes. Circ Arrhythm Electrophysiol. 2022 Aug;15(8):e010850. doi: 10.1161/CIRCEP.122.010850. Epub 2022 Jul 22. PMID 35867397
- [Background] Svennberg E, Han JK, Caiani EG, Engelhardt S, Ernst S, Friedman P, Garcia R, Ghanbari H, Hindricks G, Man SH, Millet J, Narayan SM, Ng GA, Noseworthy PA, Tjong FVY, Ramirez J, Singh JP, Trayanova N, Duncker D, Tfelt Hansen J, Barker J, Casado-Arroyo R, Chatterjee NA, Conte G, Diederichsen SZ, Linz D, Mahtani AU, Zorzi A. State of the Art of Artificial Intelligence in Clinical Electrophysiology in 2025: A Scientific Statement of the European Heart Rhythm Association (EHRA) of the ESC, the Heart Rhythm Society (HRS), and the ESC Working Group on E-Cardiology. Europace. 2025 May 7;27(5):euaf071. doi: 10.1093/europace/euaf071. PMID 40163651
- [Background] Armoundas AA, Narayan SM, Arnett DK, Spector-Bagdady K, Bennett DA, Celi LA, Friedman PA, Gollob MH, Hall JL, Kwitek AE, Lett E, Menon BK, Sheehan KA, Al-Zaiti SS; American Heart Association Institute for Precision Cardiovascular Medicine; Council on Cardiovascular and Stroke Nursing; Council on Lifelong Congenital Heart Disease and Heart Health in the Young; Council on Cardiovascular Radiology and Intervention; Council on Hypertension; Council on the Kidney in Cardiovascular Disease; and Stroke Council. Use of Artificial Intelligence in Improving Outcomes in Heart Disease: A Scientific Statement From the American Heart Association. Circulation. 2024 Apr 2;149(14):e1028-e1050. doi: 10.1161/CIR.0000000000001201. Epub 2024 Feb 28. PMID 38415358
- [Background] Narayan SM, Wan EY, Andrade JG, Avari Silva JN, Bhatia NK, Deneke T, Deshmukh AJ, Chon KH, Erickson L, Ghanbari H, Noseworthy PA, Pathak RK, Roelle L, Seiler A, Singh JP, Srivatsa UN, Trela A, Tsiperfal A, Varma N, Yousuf OK. Visions for digital integrated cardiovascular care: HRS Digital Health Committee perspectives. Cardiovasc Digit Health J. 2024 Feb 24;5(2):37-49. doi: 10.1016/j.cvdhj.2024.02.003. eCollection 2024 Apr. No abstract available. PMID 38765620
- [Background] Armoundas AA, Ahmad FS, Bennett DA, Chung MK, Davis LL, Dunn J, Narayan SM, Slotwiner DJ, Wiley KK Jr, Khera R; American Heart Association Data Science and Precision Medicine Committee of the Council on Genomic and Precision Medicine and Council on Clinical Cardiology; Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; Council on Cardiovascular and Stroke Nursing; Council on Lifestyle and Cardiometabolic Health; Council on Peripheral Vascular Disease; Council on Quality of Care and Outcomes Research; and Stroke Council. Data Interoperability for Ambulatory Monitoring of Cardiovascular Disease: A Scientific Statement From the American Heart Association. Circ Genom Precis Med. 2024 Jun;17(3):e000095. doi: 10.1161/HCG.0000000000000095. Epub 2024 May 23. PMID 38779844
- [Background] de Groot NMS, Kleber A, Narayan SM, Ciaccio EJ, Doessel O, Bernus O, Berenfeld O, Callans D, Fedorov V, Hummel J, Haissaguerre M, Natale A, Trayanova N, Spector P, Vigmond E, Anter E. Atrial fibrillation nomenclature, definitions, and mechanisms: Position paper from the international Working Group of the Signal Summit. Heart Rhythm. 2025 Jun;22(6):1480-1491. doi: 10.1016/j.hrthm.2024.11.012. Epub 2024 Nov 17. PMID 39561931
- [Background] Goldberger JJ, Mitrani RD, Zaatari G, Narayan SM. Mechanistic Insights From Trials of Atrial Fibrillation Ablation: Charting a Course for the Future. Circ Arrhythm Electrophysiol. 2024 Aug;17(8):e012939. doi: 10.1161/CIRCEP.124.012939. Epub 2024 Jul 23. PMID 39041221
- [Background] Sillett C, Razeghi O, Baptiste TMG, Lee AWC, Solis Lemus JA, Rodero C, Roney CH, Feng R, Ganesan P, Chang HJ, Clopton P, Linton N, Rajani R, Rogers AJ, Narayan SM, Niederer SA. Identification of atrial myopathy and atrial fibrillation recurrence after ablation using 3D left atrial phasic strain from retrospective gated computed tomography. Eur Heart J Imaging Methods Pract. 2025 Mar 6;3(1):qyaf027. doi: 10.1093/ehjimp/qyaf027. eCollection 2025 Jan. PMID 40171523
- [Background] Ganesan P, Deb B, Feng R, Rodrigo M, Ruiperez-Campillo S, Rogers AJ, Clopton P, Wang PJ, Zeemering S, Schotten U, Rappel WJ, Narayan SM. Quantifying a spectrum of clinical response in atrial tachyarrhythmias using spatiotemporal synchronization of electrograms. Europace. 2023 May 19;25(5):euad055. doi: 10.1093/europace/euad055. PMID 36932716
- [Background] Feng R, Deb B, Ganesan P, Tjong FVY, Rogers AJ, Ruiperez-Campillo S, Somani S, Clopton P, Baykaner T, Rodrigo M, Zou J, Haddad F, Zahari M, Narayan SM. Segmenting computed tomograms for cardiac ablation using machine learning leveraged by domain knowledge encoding. Front Cardiovasc Med. 2023 Oct 2;10:1189293. doi: 10.3389/fcvm.2023.1189293. eCollection 2023. PMID 37849936
- [Background] Ganesan P, Pedron M, Feng R, Rogers AJ, Deb B, Chang HJ, Ruiperez-Campillo S, Srivastava V, Brennan KA, Giles WR, Baykaner T, Clopton P, Wang PJ, Schotten U, Krummen DE, Narayan SM. Comparing Phenotypes for Acute and Long-Term Response to Atrial Fibrillation Ablation Using Machine Learning. Circ Arrhythm Electrophysiol. 2025 Feb;18(2):e012860. doi: 10.1161/CIRCEP.124.012860. Epub 2025 Feb 10. PMID 39925268
- [Background] Narayan SM, Krummen DE, Shivkumar K, Clopton P, Rappel WJ, Miller JM. Treatment of atrial fibrillation by the ablation of localized sources: CONFIRM (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation) trial. J Am Coll Cardiol. 2012 Aug 14;60(7):628-36. doi: 10.1016/j.jacc.2012.05.022. Epub 2012 Jul 18. PMID 22818076
- [Background] Narayan SM, Krummen DE, Enyeart MW, Rappel WJ. Computational mapping identifies localized mechanisms for ablation of atrial fibrillation. PLoS One. 2012;7(9):e46034. doi: 10.1371/journal.pone.0046034. Epub 2012 Sep 26. PMID 23049929
- [Background] Benharash P, Buch E, Frank P, Share M, Tung R, Shivkumar K, Mandapati R. Quantitative analysis of localized sources identified by focal impulse and rotor modulation mapping in atrial fibrillation. Circ Arrhythm Electrophysiol. 2015 Jun;8(3):554-61. doi: 10.1161/CIRCEP.115.002721. Epub 2015 Apr 14. PMID 25873718
- [Background] Jalife J, Filgueiras Rama D, Berenfeld O. Letter by Jalife et al Regarding Article, "Quantitative Analysis of Localized Sources Identified by Focal Impulse and Rotor Modulation Mapping in Atrial Fibrillation". Circ Arrhythm Electrophysiol. 2015 Oct;8(5):1296-8. doi: 10.1161/CIRCEP.115.003324. No abstract available. PMID 26487627
- [Background] Kuklik P, Zeemering S, Maesen B, Maessen J, Crijns HJ, Verheule S, Ganesan AN, Schotten U. Reconstruction of instantaneous phase of unipolar atrial contact electrogram using a concept of sinusoidal recomposition and Hilbert transform. IEEE Trans Biomed Eng. 2015 Jan;62(1):296-302. doi: 10.1109/TBME.2014.2350029. Epub 2014 Aug 20. PMID 25148659
- [Background] Kuklik P, Zeemering S, van Hunnik A, Maesen B, Pison L, Lau DH, Maessen J, Podziemski P, Meyer C, Schaffer B, Crijns H, Willems S, Schotten U. Identification of Rotors during Human Atrial Fibrillation Using Contact Mapping and Phase Singularity Detection: Technical Considerations. IEEE Trans Biomed Eng. 2017 Feb;64(2):310-318. doi: 10.1109/TBME.2016.2554660. Epub 2016 Apr 15. PMID 27101596
- [Background] Haissaguerre M, Hocini M, Denis A, Shah AJ, Komatsu Y, Yamashita S, Daly M, Amraoui S, Zellerhoff S, Picat MQ, Quotb A, Jesel L, Lim H, Ploux S, Bordachar P, Attuel G, Meillet V, Ritter P, Derval N, Sacher F, Bernus O, Cochet H, Jais P, Dubois R. Driver domains in persistent atrial fibrillation. Circulation. 2014 Aug 12;130(7):530-8. doi: 10.1161/CIRCULATIONAHA.113.005421. Epub 2014 Jul 15. PMID 25028391
- [Derived] Kowalewski CAB, Shenasa F, Rodrigo M, Clopton P, Meckler G, Alhusseini MI, Swerdlow MA, Joshi V, Hossainy S, Zaman JAB, Baykaner T, Rogers AJ, Brachmann J, Miller JM, Krummen DE, Sauer WH, Peters NS, Wang PJ, Narayan SM. Interaction of Localized Drivers and Disorganized Activation in Persistent Atrial Fibrillation: Reconciling Putative Mechanisms Using Multiple Mapping Techniques. Circ Arrhythm Electrophysiol. 2018 Jun;11(6):e005846. doi: 10.1161/CIRCEP.117.005846. PMID 29884620